CLINICAL TRIAL: NCT07157189
Title: Clinical, Laboratory and Therapeutic Profile of Behçet's Disease Patients in Tertiary Center in Upper Egypt
Brief Title: Clinical, Laboratory, and Therapeutic Analysis of Behçet's Disease in Assiut
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Maher, resident at the Rheumatology, Rehabilitation and Physical Medicine department, Assiut University
Other Study IDs: Analysis of Behçet's Disease
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Behçet's Disease
Keywords: Behçet's disease; therapeutic profile
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Behçet's disease patients: adults and adolescents diagnosed using international criteria (ISG and rICBD), with recurrent oral ulceration and at least two additional manifestations (genital ulcers, eye lesions, skin lesions, positive pathergy test).

SUMMARY:
A cross-sectional, observational study surveying the clinical, laboratory, and therapeutic characteristics of Behçet's disease patients in a tertiary care center in Upper Egypt

DETAILED DESCRIPTION:
This research is designed to comprehensively characterize Behçet's disease (BD), an inflammatory multisystem disorder with variable prevalence and presentation based on geography and ethnicity. Data will be collected from patients attending the Rheumatology, Rehabilitation and Physical Medicine department, Assiut University Hospitals, capturing demographic profiles, disease manifestations, laboratory results, and therapeutic history. The study uses validated criteria (ISG and rICBD) for BD diagnosis, focusing on thorough examination across musculoskeletal, dermatological, ocular, vascular, gastrointestinal, and neurological domains. Disease activity and severity will be assessed using standardized forms (Behcet's disease current activity form 2006, BODI). Laboratory analysis includes CBC, acute phase reactants, and organ function tests. Data management incorporates advanced statistical techniques using SPSS, aiming for rigorous analysis to inform future BD management in the region .

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfil the international study group criteria (ISG) which require the presence of recurrent oral ulceration plus at least two of the following: recurrent genital ulcers, eye lesions (uveitis or retinal vasculitis), skin lesions, or a positive pathergy test (12). and the revised International Criteria of BD (rICBD)

Exclusion Criteria:

* Patients with unconfirmed diagnosis of BD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are adults and adolescents diagnosed using international criteria (ISG and rICBD), with recurrent oral ulceration and at least two additional manifestations (genital ulcers, eye lesions, skin lesions, positive pathergy test). Patients with unconfirmed BD are excluded. Given BD's variable age and gender distribution, the population will reflect regional epidemiological trends, including a probable male predominance consistent with Arab and Mediterranean cohorts. Comprehensive sociodemographic data, disease duration, age at onset, family/personal history, and clinical presentation are documented. All patients are monitored through a structured two-year inclusion, maximizing sample heterogeneity and capturing real-world data from both inpatient and outpatient clinical pathways .
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-09-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of key clinical manifestations in Behçet's disease patients | Baseline
  This outcome will systematically quantify how often major clinical features-such as recurrent oral ulcers, genital ulcers, ocular lesions (including chronic relapsing uveitis), and musculoskeletal involvement, appear within the studied Behçet's disease population, in accordance with predefined diagnostic criteria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazaa A, Makhlouf Y, Ben Massoud F, Miladi S, Boussaa H, Ouenniche K, Souebni L, Kassab S, Chekili S, Ben Abdelghani K, Laatar A. Behcet disease: epidemiology, classification criteria and treatment modalities. Expert Rev Clin Immunol. 2024 Dec;20(12):1437-1448. doi: 10.1080/1744666X.2024.2388693. Epub 2024 Aug 11. PMID 39101633